CLINICAL TRIAL: NCT06077656
Title: A Phase 2, Multicenter, Randomized, Active-Controlled, Observer-Blind, Dose-Ranging Study to Evaluate the Safety, Tolerability, and Immunogenicity of a 25-Valent Pneumococcal Conjugate Vaccine in Healthy PCV-Naïve Adults
Brief Title: Dose-Ranging Study to Evaluate a 25-Valent Pneumococcal Conjugate Vaccine
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Inventprise Inc. (Industry)
Collaborators: Canadian Center for Vaccinology (Other); Vaccine Evaluation Center, Canada (Other); PATH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CVIA 105
Record Dates: First submitted 2023-10-05; First posted 2023-10-11 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Pneumococcal Vaccines

STUDY DESIGN:
Intervention Model Description: Multicenter, randomized, active-controlled, observer-blind study to evaluate safety, tolerability, and immunogenicity of three formulations of IVT PCV-25 in which healthy adult participants will be randomized in a 4:3:2:2 ratio to receive 1 of 3 formulations or control.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A (Experimental): Participants will receive a single 0.5mL dose of IVT PCV-25 Formulation A administered by intramuscular injection on Day 1
  Interventions: Biological: IVT PCV-25 Formulation A
- Group B (Experimental): Participants will receive a single 0.5mL dose of IVT PCV-25 Formulation B administered by intramuscular injection on Day 1
  Interventions: Biological: IVT PCV-25 Formulation B
- Group C (Experimental): Participants will receive a single 0.5mL dose of IVT PCV-25 Formulation C administered by intramuscular injection on Day 1
  Interventions: Biological: IVT PCV-25 Formulation C
- Group D (Active Comparator): Participants will receive a single 0.5mL dose of PCV 20 administered by intramuscular injection on Day 1
  Interventions: Biological: PCV 20

INTERVENTIONS:
Biological: IVT PCV-25 Formulation A — 25 valent pneumococcal conjugate vaccine containing low dose polysaccharide and low dose adjuvant
  Arms: Group A
Biological: IVT PCV-25 Formulation B — 25 valent pneumococcal conjugate vaccine containing low dose polysaccharide and high dose adjuvant
  Arms: Group B
Biological: IVT PCV-25 Formulation C — 25 valent pneumococcal conjugate vaccine containing high dose polysaccharide and high dose adjuvant
  Arms: Group C
Biological: PCV 20 — 20 valent pneumococcal conjugate vaccine
  Arms: Group D

SUMMARY:
Phase 2 trial to evaluate safety, tolerability, and immunogenicity of Inventprise's (IVT) 25-valent pneumococcal conjugate vaccine (IVT PCV-25)

DETAILED DESCRIPTION:
A Phase 2 multicenter, randomized, active-controlled, observer-blind study to evaluate safety, tolerability, and immunogenicity of three formulations of IVT PCV-25, a 25 valent conjugated pneumococcal vaccine with adjuvant. Adult participants will be randomized in a 4:3:2:2 ratio to receive 1 of 3 formulations or control.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults who are 18 through 49 years old on the day of randomization (Day 1).
* Participant must provide voluntary written informed consent to participate in the study.
* Participant must be able to comprehend and comply with study requirements and procedures and be willing and able to return for all scheduled follow-up visits.
* Adult female participants who are not surgically sterile must have a negative pregnancy test at screening and negative pregnancy test prior to vaccination and must agree to employ a highly effective method to avoid pregnancy through Day 57 of the study.

Exclusion Criteria:

* Use of any investigational medicinal product within 90 days prior to randomization or planned use of such a product during the period of study participation.
* Adults who have previously been vaccinated against S. pneumoniae.
* History of microbiologically confirmed invasive disease caused by S. pneumoniae.
* History of allergic disease (including angioedema) or history of a serious reaction to any prior vaccination or known hypersensitivity to any component of the study vaccines, including PEG.
* Any abnormal vital sign deemed clinically relevant by the PI.
* Acute illness at time of randomization (moderate or severe) and/or fever (body temperature of ≥ 38.0°C)
* History of any non-study vaccine administration within 14 days of study vaccine administration.
* No planned vaccines until after Day 29 (Visit 3).
* Chronic administration (defined as more than 14 consecutive days) of immunosuppressant or other immune modifying drugs prior to the administration of the study vaccine (and within the 6 months prior to administration of the study vaccine), including the use of glucocorticoids. The use of topical and inhaled glucocorticoids will be permitted.
* Administration of immunoglobulins and/or any blood products within the 6 months prior to administration of the study vaccine or anticipation of such administration during the study period.
* Any medical or social condition that in the opinion of the PI , may interfere with the study objectives, pose a risk to the participant, or prevent the participant from completing the study follow-up.
* Any screening laboratory test result outside the normal range and with toxicity score ≥ 2, unless allowed by study team.
* A positive serologic test for human immunodeficiency virus (HIV)-1 or HIV-2 (HIV 1/2 Ab), hepatitis B (HBsAg) or hepatitis C (HCV Ab).
* History of malignancy, excluding non-melanoma skin and cervical carcinoma in situ.
* Recent history (within the past year) or signs of alcohol or substance abuse.
* History of major psychiatric disorder.
* Female adult participants who are pregnant or breastfeeding.
* Participant is an employee of, or direct descendant (child or grandchild) of any person employed by the Sponsor, PATH, the Contract Research Organization (CRO), the PI.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 220 (Estimated)
Dates: Start 2023-10-25 (Actual); Primary Completion 2024-05-24 (Estimated); Study Completion 2024-05-24 (Estimated)

PRIMARY OUTCOMES:
Solicited local adverse events (AEs) | 7 days post-vaccination (Day 8)
  Number and severity of solicited local AEs
Solicited systemic AEs | 7 days post-vaccination (Day 8)
  Number and severity of solicited systemic AEs
Unsolicited AEs | 28 days post-vaccination (Day 29)
  Number and severity of unsolicited AEs
Severe adverse events (SAEs) | 6 months post-vaccination (Day 169)
  Number of SAEs

SECONDARY OUTCOMES:
Immunoglobulin G (IgG) geometric mean concentration (GMC) | Baseline (Day 1) and 28 days post-vaccination (Day 29)
  Serotype-specific IgG GMCs
IgG geometric mean fold rise (GMFR) | 28 days post-vaccination (Day 29)
  IgG GMFR as measured by serotype-specific IgG GMCs from baseline
IgG four-fold rise | 28 days post-vaccination (Day 29)
  Percentage of participants with four-fold IgG GMC rise or greater as measured by serotype-specific IgG GMCs from baseline
IgG GMC ratio | 28 days post-vaccination (Day 29)
  IgG GMC ratio between IVT PCV-25 and Prevnar 20 groups as measured by serotype-specific IgG GMCs
IgG GMFR ratio | 28 days post-vaccination (Day 29)
  IgG GMFR ratio between IVT PCV-25 and Prevnar 20 groups as measured by serotype-specific IgG GMCs
OPA geometric mean titer (GMT) | Baseline (Day 1) and 28 days post-vaccination (Day 29)
  Serotype-specific OPA GMTs
OPA GMFR | 28 days post-vaccination (Day 29)
  OPA GMFR between IVT PCV-25 and Prevnar 20 groups as measured by serotype-specific OPA GMTs from baseline
OPA GMT ratio | 28 days post-vaccination (Day 29)
  OPA GMT ratio between IVT PCV-25 and Prevnar 20 groups as measured by serotype-specific OPA GMTs
OPA GMFR ratio | 28 days post-vaccination (Day 29)
  OPA GMFR ratio between IVT PCV-25 and Prevnar 20 groups as measured by serotype-specific OPA GMTs

CONTACTS AND LOCATIONS:
Overall Officials: Sybil Tasker, MD, MPH, FIDSA, Study Director — Inventprise Inc.
Locations (4):
- Canada (4):
  - Inventprise Clinical Site, Vancouver, British Columbia
  - Inventprise Clinical Site, Halifax, Nova Scotia
  - Inventprise Clinical Site, Truro, Nova Scotia
  - Inventprise Clinical Site, Saint-Louis, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Plan to be defined at a later date
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Plan to be defined at a later date
Access Criteria: Plan to be defined at a later date

REFERENCES:
- [Derived] Langley JM, Sadarangani M, Ockenhouse C, Barreto L, Ye L, Tang Y, Breeze JL, Feser J, Hosken NA, Andi-Lolo I, Tasker SA, Halperin SA; Canadian Immunization Research Network. Safety and immunogenicity of a 25-valent pneumococcal conjugate vaccine in pneumococcal vaccine-naive healthy adults: Results from 2 randomised, controlled clinical trials. Vaccine. 2026 Jan 22;75:128236. doi: 10.1016/j.vaccine.2026.128236. Online ahead of print. PMID 41576705